CLINICAL TRIAL: NCT01475552
Title: The Effect of Point-of-care Platelet Function Assay Guided Antiplatelet Therapy on the Periprocedural Increase of Cardiac Enzymes.
Brief Title: Tailored Antiplatelet Therapy During Percutaneous Coronary Intervention in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DM-Verifynow
Record Dates: First submitted 2011-11-14; First posted 2011-11-21 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus
Keywords: platelet reactivity; platelet function assay; abciximab; tailored therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Abciximab; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- abciximab (Experimental)
  Interventions: Drug: Abciximab
- control (Active Comparator)
  Interventions: Drug: control

INTERVENTIONS:
Drug: Abciximab — Patients, who showed PRU >270 unit and were randomized to abciximab group,were treated with abciximab in addition to conventional antiplatelet treatment (aspirin+clopidogrel).
  Other Names: *Reopro, Lily Korea; Dose: 0.25mg/kg intravenous bolus injection and 0.125ug/kg/min continuous infusion for 12hrs
  Arms: abciximab
Drug: control — Patients,who showed PRU >270 unit and were randomized to control group,were treated with conventional antiplatelet therapy (aspirin+clopidogrel) during PCI and follow up periods.
  Aspirin : D-1 300mg, D0-30 100mg qd Clopidogrel : D-1 300mg, D0-30 75mg qd
  Other Names: Aspirin; Clopidogrel (Plavix)
  Arms: control

SUMMARY:
The researchers aimed to investigate the effect of point-of-care platelet function assay on the periprocedural cardiac enzyme elevation in patients with diabetes mellitus.

All patients who are supposed to undergo coronary angiography were loaded with clopidogrel (300mg) and aspirin (300mg) at D-1. If patients were determined to implant coronary stent after diagnostic coronary angiography, their platelet function is assayed with Verifynow-ADP (Accumetrics). If patients have >270 unit in the assay, they are randomized to abciximab or control group. After successful stent implantation, cardiac enzymes (CK-MB, Troponin-I) are followed at 8hr, 16hr and 24hr. Clinical outcomes including bleeding complications are assessed at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were determined to implant drug-eluting coronary stent
* Diabetes mellitus (type 1 or 2)

Exclusion Criteria:

* Age <18 years or >80years
* Patients with acute myocardial infarction
* Patients with history of cerebral hemorrhage ever or ischemic infarction within 2 years
* Patients with history of major surgery (abdominal, thoracic, intraocular) within 6 months
* Patients who have have allergy to antiplatelet medications (aspirin, clopidogrel, abciximab)
* Patients who are on anticoagulation therapy
* Serum creatinine >2.0mg/dl or ALT/AST > 3 times of upper normal limit (120 U/L)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Peak cardiac enzyme level (CK-MB,troponin-I) | within 24 hrs
  The investigators will check cardiac enzymes at 8hrs, 16hrs and 24hrs after percutaneous coronary intervention. We will take the highest value among those measured at three time points as a patient's peak cardiac enzyme level. The primary outcome of this study is to compare the peak cardiac enzyme level between two groups.

SECONDARY OUTCOMES:
major adverse cardiovascular events (MACE): a composite of cardiac death, myocardial infarction, ischemic stroke | 1 month
Bleeding complications (cerebrovascular, intraocular, bleeding which needs transfusion more than 2 pints) | 1 month
The rate of periprocedural myocardial infarction | 8hr, 16hr, 24hrs
  The definition of periprocedural myocardial infarction : cardiac enzyme increase more than three times of upper normal limit

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, MD,PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea